CLINICAL TRIAL: NCT04399733
Title: EMPOWER - BAME vs COVID: A Multi-site Clinical Cohort Research Study to Identify Genetic Associations and Candidate Therapeutic Targets to Reduce COVID-19 Morbidity & Mortality Rates in BAME Populations
Brief Title: EMPOWER - BAME vs COVID
Status: Withdrawn | Type: Observational
Why Stopped: Vaccine rollouts in UK
Sponsor: Future Genetics Limited (Other)
Responsible Party: Sponsor
Other Study IDs: EMPOWER-BAME vs COVID
Record Dates: First submitted 2020-05-21; First posted 2020-05-22 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: COVID-19, SARS-CoV 2 Infection; Health Disparities
Keywords: ethnic minority, health disparity, epidemiology, biomarker discovery, public health, BAME, morbidity, mortality, COVID-19, SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ethnicity: Patients will be segmented on a 1:1:1 ratio similar to the EMPOWER-1 study based on ethnicity (White, Black, South Asian).

SUMMARY:
The COVID-19 virus pandemic has massively affected us all. Moreover, there is a disproportionately high number of COVID-19 severe infections and deaths in British Black, Asian and minority ethnic (BAME) patients. This clinical study plans to discover new ways of protecting people from this virus by looking at our DNA and biology.

DETAILED DESCRIPTION:
The COVID-19 virus pandemic has massively affected us all. We now know there is a much larger proportion of British Black, Asian and minority ethnic (BAME) patients suffering from COVID-19 infections. This disproportionate level of infection and severity of disease has raised concerns and worries. Other research from April 2020 showed that 71% of the nurses and midwives and 94% of the doctors and dentists that died of COVID-19 infections were from a BAME background despite this group representing 20% and 44% of the workforce respectively. The survival picture is also grim for Black and Asian members of the public where we see disproportionately high rates of deaths. Research estimates that our DNA and the environment equally influence the risk for infection. This clinical study plans to better understand our DNA. Some of the things we will be looking at is age, sex, ethnicity and any illnesses such as diabetes or blood pressure. We will ask people for some spit and look at their medical records. This may help us find some of the reasons why this virus has different effects on people and how we might protect people from COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. All competent adult and children above the age of 5 years
2. Subjects agree to:

   1. Gift saliva (spit) samples
   2. Provide Consent for access to medical and health records

Exclusion Criteria:

1. Patient is not registered with the NHS for care.
2. Adults lacking capacity
3. Children under the age of 6 years.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who are registered as UK NHS patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Identify COVID-19 specific host-defence ("protective") or predisposing ("susceptibility") genetic biomarkers | 30 months
  Discovery of genetic associations with COVID-19 infections that may form the basis of prevention, treatment or management of at-risk BAME groups and the wider population.

SECONDARY OUTCOMES:
Epidemiological profiles of COVID-19 infections in different UK ethnic populations | 24 months
  Measure the variation and extent of the different types of COVID-19 infection in different populations

CONTACTS AND LOCATIONS:
Overall Officials: Dr Mohammed Kamran, Principal Investigator — Future Genetics Limited
Locations (1):
- Future Genetics Limited, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FUTURE GENETICS website — https://futuregenetics.co.uk/